CLINICAL TRIAL: NCT05029479
Title: Clinical Performance of a Moisture Resistant, M-TEG-P Phosphate Monomer-based Universal Adhesive in Geriatric Patients With Non-carious Cervical Lesions (NCLLs):A Randomized Clinical Trial
Brief Title: the Clinical Performance of a Moisture Resistant, M-TEG-P Phosphate Monomer Based Universal Adhesive (YAMAKIN TMR-Aquabond0) Compared to the Conventional Universal Adhesive (3m ESPE Single Bond Universal Adhesive)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Taha Hanafi Mahmoud, Resident in Conservative dentistry department , Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Novel YAMAKIN TMR-Aquabond0
Record Dates: First submitted 2021-08-21; First posted 2021-08-31 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Non-carious Cervical Lesions; Geriatric Patients
Keywords: Non-Carious cervical lesions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yamakin TMR-Aquabond0 (Experimental): Novel Moisture Resistant, M-TEG-P Phosphate Monomer Based Universal Adhesive (YAMAKIN TMR-Aquabond0)
  Interventions: Other: Bonding in NCCLs
- 3m ESPE Single Bond Universal Adhesive (Active Comparator): Conventional Universal Adhesive
  Interventions: Other: Bonding in NCCLs

INTERVENTIONS:
Other: Bonding in NCCLs — bonding agent which can resist moisture and has shorter decalcifying and curing time

SUMMARY:
this trial is to test the clinical performance of a novel moisture resistant, M-TEG-P phosphate monomer based universal adhesive (YAMAKIN TMR-Aquabond0) compared to the conventional universal adhesive (3m ESPE Single Bond Universal Adhesive) in geriatric patients with Non-carious Cervical lesions (NCLLs)

DETAILED DESCRIPTION:
To evaluate the clinical performance of a novel moisture resistant, M-TEG-P phosphate monomer based universal adhesive (YAMAKIN TMR-Aquabond0) compared to the conventional universal adhesive (3m ESPE Single Bond Universal Adhesive) in geriatric patients with Non-carious Cervical lesions (NCLLs)

P: Population: Geriatric patients with non-carious cervical lesions (NCCLs) I: Intervention: Novel moisture resistant, M-TEG-P phosphate monomer based universal adhesive (YAMAKIN TMR-Aquabond0) C: Comparator : 3m ESPE Single Bond Universal Adhesive O: Outcome:Clinical Performance using FDI criteria

ELIGIBILITY:
Inclusion Criteria:

1. Non-carious cervical lesions in anterior and posterior teeth.
2. Geriatric patients from age 60 years and above.
3. Patients willing to commit to the whole period of the study.
4. Males & Females included.

Exclusion Criteria:

1. Lack of written informed consent to participate
2. Cervical hypersensitivities
3. Underage patients
4. Allergies to components of the materials used
5. Infectious diseases
6. Mucosal diseases with unclear diagnosis
7. Inadequate oral hygiene
8. Bruxism
9. High caries activity
10. Non-vital pulp
11. Severe periodontal diseases
12. Severe dysgnathia/traumatic occlusion
13. Undergoing orthodontic treatments
14. Undergoing bleaching procedures

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-10-13 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of fractured restorations | 12 months
  First, visual inspection to ensure that there is no complete loss of retention of the restoration then tactile evaluation will be done using probe tip that will be held gently at right angle to the labial surface and move from restoration to tooth and vice versa to insure there is no rocking /fracture /ditching in the restoration following FDI criteria ( first visually for total loss followed by tactile inspection using FDI probe for any fracture /rocking or loss of retention.
Number of restorations with retention loss | 12 months
  First, visual inspection to ensure that there is no complete loss of retention of the restoration then tactile evaluation will be done using probe tip that will be held gently at right angle to the labial surface and move from restoration to tooth and vice versa to insure no rocking /fracture /ditching in the restoration following FDI criteria

SECONDARY OUTCOMES:
Number of restoration with change in colour or texture | 12 months
  Evaluation will be done visually following FDI criteria to ensure no change in colour or texture of the restoration
Number of restoration caused biological harm | 12 months
  Evaluation will be done following FDI criteria using FDI probe to ensure there is no change in restoration that caused any harm to the health of biological structure

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li Y, Hu X, Xia Y, Ji Y, Ruan J, Weir MD, Lin X, Nie Z, Gu N, Masri R, Chang X, Xu HHK. Novel magnetic nanoparticle-containing adhesive with greater dentin bond strength and antibacterial and remineralizing capabilities. Dent Mater. 2018 Sep;34(9):1310-1322. doi: 10.1016/j.dental.2018.06.001. Epub 2018 Jun 21. PMID 29935766
- [Result] Wawrzynkiewicz A, Rozpedek-Kaminska W, Galita G, Lukomska-Szymanska M, Lapinska B, Sokolowski J, Majsterek I. The Cytotoxicity and Genotoxicity of Three Dental Universal Adhesives-An In Vitro Study. Int J Mol Sci. 2020 May 31;21(11):3950. doi: 10.3390/ijms21113950. PMID 32486393
- [Result] Santis LR, Silva TM, Haddad BA, Goncalves LL, Goncalves SE. Influence of dentin thickness on intrapulpal temperature under simulated pulpal pressure during Nd:YAG laser irradiation. Lasers Med Sci. 2017 Jan;32(1):161-167. doi: 10.1007/s10103-016-2098-1. Epub 2016 Oct 24. PMID 27778115
- [Result] Akarsu S, Karademir SA, Ertas E, Atasoy S. The effect of diode laser application on restoration of non carious cervical lesion: Clinical follow up. Niger J Clin Pract. 2020 Feb;23(2):165-171. doi: 10.4103/njcp.njcp_399_19. PMID 32031090
- [Result] Peumans M, Politano G, Van Meerbeek B. Treatment of noncarious cervical lesions: when, why, and how. Int J Esthet Dent. 2020;15(1):16-42. PMID 31994534
- [Result] Wagner A, Wendler M, Petschelt A, Belli R, Lohbauer U. Bonding performance of universal adhesives in different etching modes. J Dent. 2014 Jul;42(7):800-7. doi: 10.1016/j.jdent.2014.04.012. Epub 2014 May 6. PMID 24814138
- [Result] Ranjitha GR, Vikram R, Meena N, Vijayalakshmi L, Murthy CS. Clinical efficacy of universal adhesives for the restoration of noncarious cervical lesions: A randomized clinical trial. J Conserv Dent. 2020 May-Jun;23(3):227-232. doi: 10.4103/JCD.JCD_51_20. Epub 2020 Dec 4. PMID 33551590
- [Result] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997
- [Result] Loguercio AD, Luque-Martinez IV, Fuentes S, Reis A, Munoz MA. Effect of dentin roughness on the adhesive performance in non-carious cervical lesions: A double-blind randomized clinical trial. J Dent. 2018 Feb;69:60-69. doi: 10.1016/j.jdent.2017.09.011. Epub 2017 Sep 27. PMID 28962842
- [Result] Milia E, Cumbo E, Cardoso RJ, Gallina G. Current dental adhesives systems. A narrative review. Curr Pharm Des. 2012;18(34):5542-52. doi: 10.2174/138161212803307491. PMID 22632386
- [Result] Sawlani K, Lawson NC, Burgess JO, Lemons JE, Kinderknecht KE, Givan DA, Ramp L. Factors influencing the progression of noncarious cervical lesions: A 5-year prospective clinical evaluation. J Prosthet Dent. 2016 May;115(5):571-7. doi: 10.1016/j.prosdent.2015.10.021. Epub 2016 Jan 7. PMID 26774320
- [Result] de Paris Matos T, Perdigao J, de Paula E, Coppla F, Hass V, Scheffer RF, Reis A, Loguercio AD. Five-year clinical evaluation of a universal adhesive: A randomized double-blind trial. Dent Mater. 2020 Nov;36(11):1474-1485. doi: 10.1016/j.dental.2020.08.007. Epub 2020 Sep 12. PMID 32933775
- [Result] Luque-Martinez IV, Perdigao J, Munoz MA, Sezinando A, Reis A, Loguercio AD. Effects of solvent evaporation time on immediate adhesive properties of universal adhesives to dentin. Dent Mater. 2014 Oct;30(10):1126-35. doi: 10.1016/j.dental.2014.07.002. Epub 2014 Aug 16. PMID 25139815